CLINICAL TRIAL: NCT03961971
Title: A Phase I Trial of Anti-Tim-3 in Combination With Anti-PD-1 and SRS in Recurrent GBM
Brief Title: Trial of Anti-Tim-3 in Combination With Anti-PD-1 and SRS in Recurrent GBM
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins (Other)
Collaborators: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: J18150; IRB00104226 (Other: JHM IRB)
Record Dates: First submitted 2019-05-15; First posted 2019-05-23 (Actual); Last update posted 2025-09-10 (Actual); Status verified 2025-09

CONDITIONS: Glioblastoma Multiforme
Keywords: Immunotherapy
MeSH Terms: conditions — Glioblastoma | interventions — sabatolimab; spartalizumab; Radiosurgery

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (MBG453, spartalizumab, stereotactic radiosurgery) (Experimental): Patients receive MBG453 and spartalizumab IV over 30 minutes on Day 1. Patients then undergo stereotactic radiosurgery on Day 8. Courses with MBG453 and spartalizumab repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: MBG453

INTERVENTIONS:
Drug: MBG453 — Patients receive MBG453 and spartalizumab IV over 30 minutes on Day 1. Patients then undergo stereotactic radiosurgery on Day 8. Courses with MBG453 and spartalizumab repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  Other Names: spartalizumab; stereotactic radiosurgery

SUMMARY:
This phase I trial studies the side effects of stereotactic radiosurgery with MBG453 and spartalizumab in treating patients with recurrent glioblastoma multiforme (GBM). Stereotactic radiosurgery is a specialized radiation therapy that delivers a single, high dose of radiation directly to the tumor to more precisely target the cancer. Monoclonal antibodies, such as MBG453 and spartalizumab may interfere with the ability of tumor cells to grow and spread. Giving stereotactic radiosurgery together with immunotherapy may be a better treatment for GBM.

DETAILED DESCRIPTION:
Primary Objectives To determine safety of MBG453 given in combination with spartalizumab and SRS in patients with recurrent GBM.

Secondary Objectives

To assess the preliminary anti-tumor activity using the following measures:

1. To estimate overall survival
2. To estimate progression-free survival
3. To estimate Radiographic Response (RANO and iRANO)
4. To evaluate pain for patients undergoing the treatment of anti-TIM3 and anti-PD1 in combination with SRS

Exploratory Objectives

1. To assess the effects of MGB453, spartalizumab and their combination with SRS on immune cells in peripheral blood, including but not limited to the T cell compartments, myeloid cells, and serum proteins (cytokines and other immune modulators).
2. To assess the pharmacodynamic activity in tumor tissue and peripheral blood in treated subjects who undergo tumor biopsies as clinically indicated.
3. To explore potential associations between biomarker measures and anti-tumor activity by analyzing markers of inflammation, immune activation, host tumor growth factors, and tumor-derived proteins in the pre-treatment and on-treatment setting.
4. To explore characteristics of tumor immune microenvironment change after the treatment.

OUTLINE:

Patients receive MBG453 and spartalizumab intravenously (IV) over 30 minutes each on Day 1. Patients then undergo stereotactic radiosurgery on Day 8 per standard of care. Courses with MBG453 and spartalizumab repeat every 28 days in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up every 3 months thereafter.

ELIGIBILITY:
Inclusion Criteria:

1. Patients must provide written informed consent prior to any screening procedures.
2. Age 18 years or older.
3. Willing and able to comply with scheduled visits, treatment plan and laboratory tests
4. Must have WHO Grade IV Glioblastoma or gliosarcoma based on histopathological OR molecular criteria
5. Patients tumor target (GTV) should be ≤ 5 cm.
6. a) Must have received first-line multimodal therapy with surgery (resection or biopsy) followed by radiation and Temozolomide (unless known MGMT promoter unmethylated) AND b) Must have completed at least 21 days of combination and Temozolomide therapy (unless known MGMT promoter unmethylated. . An interval of at least 12 weeks after the end of combination radiation therapy + Temozolomide is required unless there is: i.) Histopathologic confirmation of recurrent tumor, or ii) new enhancement on MRI outside of the radiotherapy treatment field. (*NOTE: Patients treated with Optune device or who received Gliadel wafers placed during the first surgery are eligible.
7. Must have no more than 2 recurrences of either GBM or gliosarcoma. Recurrence must be confirmed by diagnostic biopsy/surgery with local pathology review OR contrast-enhanced MRI measurable by RANO criteria. (*NOTE: Patients diagnosed with WHO Grade III that undergo surgical resection and are found to have WHO Grade IV or gliosarcoma are considered eligible).
8. Prior gamma knife, stereotactic radiosurgery, or other focal high-dose radiotherapy is allowed but the subject must have either histopathologic confirmation of recurrent tumor, or new enhancement on MRI outside of the radiotherapy treatment field
9. Karnofsky Performance Status ≥ 70
10. Must have ability to undergo MRI scans
11. Must be > 30 days since last chemotherapy
12. Must have recovered from severe toxicity of prior therapy. (NOTE: Patients who undergo surgical resection must have recovered from surgery (at least 2 weeks) before starting study treatment).
13. Subjects must have normal organ and marrow function as defined below:

    WBC ≥ 2,000/mcL absolute neutrophil count ≥ 1,500/mcL platelets ≥ 100,000/mcL hemoglobin ≥ 9.0 g/dL lymphocytes ≥ 500/mcL total bilirubin ≤ 1.5X institutional upper limit of normal AST/ALT ≤ 3.0 X institutional upper limit of normal creatinine ≤ 1.5X institutional upper limit of normal OR Creatinine clearance (CrCl) ≥ 50 mL/min (using the Cockcroft-Gault formula)
14. Women of childbearing potential (WOCBP) must have a negative serum or urine pregnancy test within -7 days prior to the start of therapy. Women must not be breastfeeding.
15. Women of child bearing potential (WOCBP) and men must use a reliable form of contraception during the study treatment period and for 150 days following the last dose of study drug. In order for a woman to be determined not of child-bearing potential, she must have ≥ 12 months of non-therapy-induced amenorrhea or be surgically sterile.

Exclusion Criteria:

1. History of other malignancy, unless the patient has been disease-free for at ≥5 years. Curatively treated basal or squamous cell carcinoma of the skin, totally excised melanoma of stage IIA or lower, low or intermediate-grade localized prostate cancer (Gleason sum ≤7), and curatively-treated carcinoma in situ of the cervix, breast, or bladder are allowed regardless.
2. Any known metastatic extracranial or leptomeningeal disease.
3. Evidence of acute intracranial / intra-tumoral hemorrhage
4. History of organ or hematopoietic stem cell (HSC) transplant
5. Receiving greater than 4 mg dexamethasone/day (or equivalent amount of an alternative corticosteroid) for a minimum of 5 days prior to screening visit. Subjects with an autoimmune condition requiring systemic treatment with either corticosteroids (> 10 mg daily prednisone or equivalent) or other immunosuppressive medications within 14 days of study entry *NOTE: Inhaled or topical steroids, and adrenal replacement steroid doses > 10 mg daily prednisone or equivalent, are permitted in the absence of active autoimmune disease
6. Prior treatment with immune-modulating therapy, other than steroids.
7. Pregnant or nursing (lactating) women
8. Known positive history of HIV, active Hepatitis B, and/or active Hepatitis C infection.
9. Subjects with active, or recent history of known or suspected autoimmune disease. Subjects with Type 1 diabetes mellitus, hypothyroidism only requiring hormone replacement, skin disorders (such as vitiligo, psoriasis, or alopecia) not requiring systemic treatment, or conditions not expected to recur in the absence of an external trigger are permitted to enroll
10. Major surgery, outside of a craniotomy/resection, within 2 weeks of the first dose of study treatment (mediastinoscopy, insertion of a central venous access device, and insertion of a feeding tube are not considered major surgery).
11. Use of any vaccines against infectious diseases (e.g. varicella, pneumococcus) within 4 weeks of initiation of study treatment
12. Any serious or uncontrolled medical disorder that, in the opinion of the investigator, may increase the risk associated with study participation or study drug administration, impair the ability of the subject to receive protocol therapy, or interfere with the interpretation of study results.
13. Subjects with interstitial lung disease that is symptomatic or may interfere with the detection or management of suspected drug-related pulmonary toxicity
14. History of evidence upon physical/neurological examination of other central nervous system condition (i.e. seizures, abscess) unrelated to cancer, unless adequately controlled by medication or considered not potentially interfering with protocol treatment.
15. History of allergy or hypersensitivity to study drug components.
16. Prisoners or subjects who are involuntarily incarcerated.
17. Subjects who are compulsorily detained for treatment of either a psychiatric or physical (e.g. infections disease) illness.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2020-02-18 (Actual); Primary Completion 2022-11-16 (Actual); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
Number of participants with serious adverse events (SAE) graded according to the National Cancer Institute Common Toxicity Criteria (NCI CTC) version 5.0 | Up to 12 weeks after first dose of study treatment
  Number of participants experiencing SAEs, as defined by NCI CTC v5.0

SECONDARY OUTCOMES:
Proportion of participants who experience grade 3 or higher toxicity, graded according to the NCI CTC v5.0 | Up to 100 days after completion of study treatment
  Proportion of participants who experience grade 3 or higher toxicity, graded according to the NCI CTC v5.0
Progression-free survival | From the date of initial diagnosis (at surgery) until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 24 months
  Progression-free survival estimated using the Kaplan-Meier method. Progression as defined by Response Assessment in Neuro-oncology (RANO) criteria: Complete Response (CR)= no change in size of T1-gadolinium-enhancing (T1-Gd+) disease, stable or reduced T2/FLAIR signal, no new lesion, no corticosteroid use, and stable or improved clinical status; Partial Response (PR)= ≥50% change in size of T1-Gd+ disease, stable or reduced T2/FLAIR signal, no new lesion, stable or reduced corticosteroid use, and stable or improved clinical status; Stable Disease (SD)= <50% reduction to <25% increase size of T1-Gd+ disease, stable or reduced T2/FLAIR signal, no new lesion, stable or reduced corticosteroid use, and stable or improved clinical status; Progressive Disease (PD)= ≥25% increase size of T1-Gd+ disease, or increased T2/FLAIR signal, or presence of new lesion, or worsening clinical status.
Overall survival | From the date of initial diagnosis until the date of death from any cause assessed up to 24 months
  Overall survival as estimated using the Kaplan-Meier method.
Objective Response | From date of baseline scan until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 24 months
  Proportion of participants who have objective PR or CR during the course of treatment and a measurable disease indicated in baseline scan. Progression is defined by Response Assessment in Neuro-oncology (RANO) criteria: Complete Response (CR)= no change in size of T1-gadolinium-enhancing (T1-Gd+) disease, stable or reduced T2/FLAIR signal, no new lesion, no corticosteroid use, and stable or improved clinical status; Partial Response (PR)= ≥50% change in size of T1-Gd+ disease, stable or reduced T2/FLAIR signal, no new lesion, stable or reduced corticosteroid use, and stable or improved clinical status; Stable Disease (SD)= <50% reduction to <25% increase size of T1-Gd+ disease, stable or reduced T2/FLAIR signal, no new lesion, stable or reduced corticosteroid use, and stable or improved clinical status; Progressive Disease (PD)= ≥25% increase size of T1-Gd+ disease, or increased T2/FLAIR signal, or presence of new lesion, or worsening clinical status.

CONTACTS AND LOCATIONS:
Overall Officials: Lawrence Kleinberg, MD, Principal Investigator — Johns Hopkins University/Sidney Kimmel Cancer Center
Locations (2):
- United States (2):
  - Stanford University, Stanford, California
  - Johns Hopkins University/Sidney Kimmel Cancer Center, Baltimore, Maryland

IPD SHARING:
Plan to Share IPD: No